CLINICAL TRIAL: NCT06397079
Title: Investigation of Effect on Oral Care Program for Residents in Long-term Care Facility
Brief Title: Oral Care Program for Residients in Long-term Care Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTH-113-3-5-004
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2024-09

CONDITIONS: Elder; Oral Hygiene
Keywords: elder; oral hygiene; long-term care facility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric toothbrush (Experimental): Teach Bass brushing technique and use electric toothbrush
  Interventions: Behavioral: Electric toothbrush
- Soft bristle toothbrush (Active Comparator): Teach Bass brushing technique and use soft bristle toothbrush
  Interventions: Behavioral: Soft bristle toothbrush

INTERVENTIONS:
Behavioral: Electric toothbrush — Teach Bass brushing technique and bursh teeth using electric toothbrush dental hygiene three times a day.
  Arms: Electric toothbrush
Behavioral: Soft bristle toothbrush — Teach Bass brushing technique and bursh teeth using soft bristle toothbrush dental hygiene three times a day.
  Arms: Soft bristle toothbrush

SUMMARY:
The aim of this study is to investigate the effectiveness of an oral care program on the oral hygiene for residents in long-term care facility.

DETAILED DESCRIPTION:
The study adopts a randomized clinical trial design and utilizes a cross-over design. The main outcomes include assessments of oral health (Oral Health Assessment Tool, Oral Health Impact Profile, Geriatric Oral Health Assessment Index), tongue coating cleanliness (Tongue Coating Index), dental plaque and gum cleanliness (Plaque Index, Gingival Index, Gingival Bleeding Index), and swallowing ability (Eating Assessment Tool, Function Oral Intake Scale, International Dysphagia Diet Standardisation Initiative).

ELIGIBILITY:
Inclusion Criteria:

1. Eating by mouth
2. Able to express fluently in Chinese after correcting vision and hearing
3. Normal hand functions
4. Able to follow instructions
5. Willing to participate in the study and sign the informed consent

Exclusion Criteria:

1. Unconsicous
2. Diagnosis of dementia and inability to communicate
3. Having a tracheostomy tube and nasogastric tube
4. Unable to move both upper limbs
5. Bedridden
6. Vulnerable populations (e.g., political, economic, or socially disadvantaged groups)

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Oral Health Assessment Tool | Baseline to 4 weeks
  The Oral Health Assessment Tool is a scale for evaluating oral health. The score ranges is 0 to 16. A higher score indicates a poorer oral health condition.
Oral Health Impact Profile | Baseline to 4 weeks
  The Oral Health Impact Profile assesses the quality of oral health-related life. The score ranges is 0 to 56. A higher score indicates poorer oral health-related quality of life.
Geriatric Oral Health Assessment Index | Baseline to 4 weeks
  The Geriatric Oral Health Assessment Index evaluates oral health for older people. The score ranges is 12 to 60. A higher score indicates better oral health.
Tongue Coating Index | Baseline to 4 weeks
  The Tongue Coating Index assesses tongue cleanliness. The score ranges is 0 to 18. A higher core indicates lower cleanliness of the tongue.
Plaque Index | Baseline to 4 weeks
  Plaque Index assesses amount of dental plaque. The score ranges is 0 to 3. A higher score indicates lower amount of dental plaque.
Gingival Index | Baseline to 4 weeks
  The Gingival Index assesses gingival health. The score ranges is 0 to 3. A higher score indicates poorer gingival health.
Gingival Bleeding Index | Baseline to 4 weeks
  The Gingival Bleeding Index assesses gingival health. The score ranges is 0 to 1. A higher score indicates poorer gingival health.
Eating Assessment Tool | Baseline to 4 weeks
  The Eating Assessment Tool evaluates the degree of swallowing status. The score ranges is 0 to 40. A higher score indicates lower swallowing ability.
Function Oral lntake Scale | Baseline to 4 weeks
  The Functional Oral Intake Scale assesses swallowing ability. The score ranges is 1 to 7. A higher score indicates greater swallowing ability.
International Dysphagia Diet Standardisation Initiative | Baseline to 4 weeks
  The International Dysphagia Diet Standardisation Initiative assesses swallowing ability. The score ranges is 0 to 7. A higher score indicates greater swallowing ability.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Xindian Dist, Taiwan